CLINICAL TRIAL: NCT02897076
Title: Dose Reduction of Antenatal Betamethasone Given to Prevent the Neonatal Complications Associated With Very Preterm Birth: a Randomized, Multicentre, Double Blind Placebo-controlled Non Inferiority Trial
Brief Title: Dose Reduction of Antenatal Betamethasone Given to Prevent the Neonatal Complications Associated With Very Preterm Birth
Acronym: BETADOSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P150944
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2020-04

CONDITIONS: Neonatal Complications
MeSH Terms: interventions — Betamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 12mg betamethasone+12mg betamethasone (Active Comparator): A betamethasone course consists in 2 intramuscular injections of 12 mg betamethasone 24 hours apart for a total dose of 24 mg.
  In the BETADOSE trial, the first injection will be unmasked in both groups. In both groups, women will received a first 12 mg injection of betamethasone according to local protocols.
  Randomization will be performed after the first injection. Women will then received either a blinded placebo injection (50% reduced dose regimen, 12 mg only from the first injection) or a second blinded 12 mg betamethasone injection (standard full dose regimen, 12 mg from the first injection and 12 mg from the second injection=24 mg).
  Interventions: Drug: betamethasone 24 mg
- 12 mg betamethasone+ placebo (Placebo Comparator): A betamethasone course consists in 2 intramuscular injections of 12 mg betamethasone 24 hours apart for a total dose of 24 mg.
  In the BETADOSE trial, the first injection will be unmasked in both groups. In both groups, women will received a first 12 mg injection of betamethasone according to local protocols.
  Randomization will be performed after the first injection. Women will then received either a blinded placebo injection (50% reduced dose regimen, 12 mg only from the first injection) or a second blinded 12 mg betamethasone injection (standard full dose regimen, 12 mg from the first injection and 12 mg from the second injection=24 mg).
  Interventions: Drug: 12mg betamethasone +placebo

INTERVENTIONS:
Drug: betamethasone 24 mg
  Arms: 12mg betamethasone+12mg betamethasone
Drug: 12mg betamethasone +placebo
  Arms: 12 mg betamethasone+ placebo

SUMMARY:
Extensive animal studies have indicated that antenatal betamethasone exposure results in altered developmental trajectories of several fetal systems. Follow up of a randomized controlled trial has shown that antenatal betamethasone exposure might result in insulin resistance 30 years later. Furthermore, animal studies and randomized trials in Humans have clearly demonstrated that betamethasone-induced growth alterations were dose-related.

In ewes, a 50% reduced dose regimen resulted in maximal improvement in preterm lamb lung function, similar to those obtained after a full dose.

Our hypothesis is that antenatal betamethasone after a 50% dose reduction, justified by the potential long term effects of this drug, is not inferior to a full dose to promote fetal lung maturation in Humans.

DETAILED DESCRIPTION:
The BETADOSE project consist in a randomized, multicenter, double blind placebo-controlled non inferiority trial comparing a standard dose regimen (24 mg) to a reduced dose regimen (12 mg) of betamethasone given to prevent the neonatal complications associated with very preterm birth.A betamethasone course consists in 2 injections of 12 mg betamethasone 24 hours apart for a total dose of 24 mg.

The first injection will be unmasked in both group. In both group, women will receive a first 12 mg injection of betamethasone according to local protocols.

Randomization will be performed after the first injection. Women will then receive either a placebo injection (reduced dose regimen, 12 mg only from the first injection) or a second 12 mg betamethasone injection (standard dose regimen, 12 mg from the first injection and 12 mg from the second injection=24 mg). This protocol allows women sent from level 1 and 2 to level 3 perinatal centers after having already received their first injection to participate.

In case of multiple antenatal betamethasone courses, women will receive their second course according to the same design as in their first course.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Patient Having receipt the first injection of betamethasone and pregnancy term < 32 weeks of gestation
* Age > 18 years
* Patient affiliated to a social security regime

Exclusion Criteria:

* Chromosomal aberrations and major fetal malformations
* Cervical dilatation ≥ 4 cm and of cervical length ≥20mm.
* Patient who have already received a first course of betamethasone
* first intravenous injection of betamethasone

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3250 (Actual)
Dates: Start 2017-01; Primary Completion 2020-01-05 (Actual); Study Completion 2020-01-05 (Actual)

PRIMARY OUTCOMES:
severe RDS defined as need for exogenous intra-tracheal surfactant in the first 48 hours of life | 48 hours of life
  The primary assessment criterion is severe respiratory distress syndrome(RDS) defined as need for exogenous intra-tracheal surfactant in the first 48 hours of life. It is considered as a binary endpoint: failure if there is occurrence of RDS, or not failure.

SECONDARY OUTCOMES:
highest appropriate fractional inspired oxygen (FiO2) | 48 hours of life
maximum appropriate Mean Airway Pressure (MAP) | 48 hours of life
duration of mechanical ventilation | 36 weeks post conception
duration of oxygen therapy | 36 weeks post conception
oxygen therapy | 36 weeks post conception
neonatal death | 36 weeks post conception
admission to neonatal intensive care unit | 36 weeks post conception
inotropic support | 36 weeks post conception
air leak syndrome | 36 weeks post conception
patent ductus arteriosus | 36 weeks post conception
necrotising enterocolitis | 36 weeks post conception
intraventricular hemorrhage and grade | 36 weeks post conception
periventricular leukomalacia | 36 weeks post conception
use of postnatal steroids | 36 weeks post conception
retinopathy of prematurity | 36 weeks post conception
length of hospital stay | 36 weeks post conception
early onset sepsis | 36 weeks post conception
Composite endpoint of any of the 4 prematurity-induced complications related to the use of betamethasone | 36 weeks post conception
  Related to betamethasone impact on other prematurity-induced complications, is a composite outcome taking into account multiple clinical events :
  neonatal death, severe RDS defined as need for exogenous intra-tracheal surfactant in the first 48 hours of life, intraventricular hemorrhage high grade, and necrotising enterocolitis.

CONTACTS AND LOCATIONS:
Overall Officials: Schmitz Thomas, PHD, Principal Investigator — APHP; Baud Olivier, PHD, Study Chair — Hôpitaux Universitaires de Genève - Inserm U1141 Hôpital Robert Debré
Locations (1):
- Hôpital Robert Debré, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmitz T, Alberti C, Ursino M, Baud O, Aupiais C; BETADOSE study group and the GROG (Groupe de Recherche en Gynecologie Obstetrique). Full versus half dose of antenatal betamethasone to prevent severe neonatal respiratory distress syndrome associated with preterm birth: study protocol for a randomised, multicenter, double blind, placebo-controlled, non-inferiority trial (BETADOSE). BMC Pregnancy Childbirth. 2019 Feb 12;19(1):67. doi: 10.1186/s12884-019-2206-x. PMID 30755164
- [Background] Aupiais C, Alberti C, Schmitz T, Baud O, Ursino M, Zohar S. A Bayesian non-inferiority approach using experts' margin elicitation - application to the monitoring of safety events. BMC Med Res Methodol. 2019 Sep 18;19(1):187. doi: 10.1186/s12874-019-0826-5. PMID 31533631
- [Result] Schmitz T, Doret-Dion M, Sentilhes L, Parant O, Claris O, Renesme L, Abbal J, Girault A, Torchin H, Houllier M, Le Sache N, Vivanti AJ, De Luca D, Winer N, Flamant C, Thuillier C, Boileau P, Blanc J, Brevaut V, Bouet PE, Gascoin G, Beucher G, Datin-Dorriere V, Bounan S, Bolot P, Poncelet C, Alberti C, Ursino M, Aupiais C, Baud O; BETADOSE trial study group; Groupe de Recherche en Obstetrique et Gynecologie. Neonatal outcomes for women at risk of preterm delivery given half dose versus full dose of antenatal betamethasone: a randomised, multicentre, double-blind, placebo-controlled, non-inferiority trial. Lancet. 2022 Aug 20;400(10352):592-604. doi: 10.1016/S0140-6736(22)01535-5. PMID 35988568